CLINICAL TRIAL: NCT03403790
Title: Drug Use-results Survey on Quetiapine Extended-release Tablets in Patients With Depression in Bipolar Disorder
Brief Title: A Survey on Quetiapine Extended-release Tablets in Patients With Depression in Bipolar Disorder
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 6949-MA-3199
Record Dates: First submitted 2018-01-07; First posted 2018-01-19 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2020-04

CONDITIONS: Depression; Bipolar Disorder
Keywords: Bipresso; Drug use-results survey; Quetiapine
MeSH Terms: conditions — Depression; Bipolar Disorder | interventions — Quetiapine Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with depression in bipolar disorder: Patients with depression in bipolar disorder who are treated with quetiapine extended-release tablets for the first time
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Quetiapine — Oral (extended-release tablet)
  Other Names: Bipresso

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of quetiapine in actual clinical settings.

DETAILED DESCRIPTION:
This is a post-marketing use-result survey study required for products in Japan. The investigator will register the patient who have been taking this product for the first time within 14 days after the start of treatment (inclusive of the start day). For each of the registered patients (including withdrawals and dropouts), the investigator will enter the survey data on the case report form.

ELIGIBILITY:
Inclusion Criteria:

* Patients with depressive symptoms of bipolar disorder
* Patients who have previously not been treated with quetiapine fumarate (immediate-release formulations of quetiapine fumarate and Bipresso Extended-Release Tablets)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with depressive symptoms of bipolar disorder who have not been treated with quetiapine fumarate
Sampling Method: Non-Probability Sample
Enrollment: 369 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Safety assessed by incidence of serious adverse events | Up to Week 12
  To assess incidence of serious adverse events as a criteria of safety variables.
Safety assessed by incidence of adverse drug reactions | Up to Week 12
  To assess incidence of adverse drug reactions as a criteria of safety variables.
Safety assessed by laboratory values and changes from baseline over time | Up to Week 12
  To assess profile of laboratory value transition and potential clinical significance as a criteria of safety variables. The investigators will assess the severity and clinical relevance, and will report as an adverse event as necessary.
Safety assessed by vital signs: Blood pressure (sitting) | Up to Week 12
  To assess blood pressure as a criteria of safety variables
Safety assessed by vital signs: Pulse rate (sitting) | Up to Week 12
  To assess pulse rate as a criteria of safety variables
Safety assessed by 12-lead electrocardiogram | Up to Week 12
  To assess 12-lead electrocardiogram as a criteria of safety variables
Safety assessed by body weight | Up to Week 12
  To assess body weight as a criteria of safety variables
Change from baseline in Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline and up to Week 12
  To assess MADRS as a criteria of efficacy variables
Change from baseline in Clinical Global Impression-Bipolar-Severity of illness (CGI-BP-S) | Baseline and up to Week 12
  To assess CGI-BP-S as a criteria of efficacy variables
Efficacy assessed by Clinical Global Impression-Bipolar-Change (CGI-BP-C) | Up to Week 12
  To assess CGI-BP-C as a criteria of efficacy variables

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Inc
Locations (47):
- Japan (47):
  - Site JP00023, Aichi
  - Site JP00005, Akita
  - Site JP00002, Aomori
  - Site JP00012, Chiba
  - Site JP00038, Ehime
  - Site JP00018, Fukui
  - Site JP00040, Fukuoka
  - Site JP00007, Fukushima
  - Site JP00021, Gifu
  - Site JP00010, Gunma
  - Site JP00034, Hiroshima
  - Site JP00001, Hokkaido
  - Site JP00028, Hyōgo
  - Site JP00008, Ibaraki
  - Site JP00017, Ishikawa
  - Site JP00037, Kagawa
  - Site JP00046, Kagoshima
  - Site JP00014, Kanagawa
  - Site JP00039, Kochi
  - Site JP00043, Kumamoto
  - Site JP00026, Kyoto
  - Site JP00024, Mie
  - Site JP00004, Miyagi
  - Site JP00045, Miyazaki
  - Site JP00020, Nagano
  - Site JP00042, Nagasaki
  - Site JP00029, Nara
  - Site JP00015, Niigata
  - Site JP00003, Numakunai
  - Site JP00033, Okayama
  - Site JP00047, Okinawa
  - Site JP00027, Osaka
  - Site JP00044, Ōita
  - Site JP00041, Saga
  - Site JP00011, Saitama
  - Site JP00025, Shiga
  - Site JP00032, Shimane
  - Site JP00022, Shizuoka
  - Site JP00009, Tochigi
  - Site JP00036, Tokushima
  - Site JP00013, Tokyo
  - Site JP00031, Tottori
  - Site JP00016, Toyama
  - Site JP00030, Wakayama
  - Site JP00006, Yamagata
  - Site JP00035, Yamaguchi
  - Site JP00019, Yamanashi

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.